CLINICAL TRIAL: NCT01398956
Title: An Open-label, Multicenter, Long-term, Follow-up Study in Japan to Evaluate the Safety, Tolerability, and Efficacy of Adjunctive Treatment With Oral L059 (Levetiracetam) in Epilepsy Subjects With Generalized Tonic-clonic (GTC) Seizures
Brief Title: An Open Label Study of L059 (Levetiracetam) in Japanese Epilepsy Subjects With Generalized Tonic-clonic Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01361
Record Dates: First submitted 2011-07-13; First posted 2011-07-21 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy; Generalized Tonic-clonic Seizures
Keywords: Levetiracetam; Epilepsy; Generalized tonic-clonic seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental): Twice daily (morning and evening) orally
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — formulation: tablet or dry syrup
  strength: 250 mg tablet, 500 mg tablet, dry syrup 50%
  dosage: Sb ≥16 years and ≥4 and <16 years (≥50 kg): 1000 mg/day, 2000 mg/day or 3000 mg/day; Sb ≥4 and <16 years (<50kg): 20 mg/kg/day, 40 mg/kg/day, or 60 mg/kg/day
  frequency: twice daily
  Other Names: Keppra, E Keppra

SUMMARY:
The investigators will provide Levetiracetam treatment to epilepsy subjects in Japan who are judged to benefit from continued treatment with Levetiracetam by the investigators and who are willing to continuously receive this drug.

ELIGIBILITY:
Inclusion Criteria:

* The subject in Japan has completed either of the studies N01159 or N01363 or has discontinued the N01159 study due to lack of efficacy.
* The subject who is judged to benefit from continued treatment with Levetiracetam by the investigators

Exclusion Criteria:

* Subjects with multiple protocol deviations during N01159 or N01363, such as missing laboratory data, and low or noncompliance with the study medication, and who the investigator considers not to have the potential to have deviations stopped are ineligible

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (32):
- Japan (32):
  - 152, Fujisawa
  - 112, Fukuoka
  - 113, Fukuoka
  - 165, Fukuoka
  - 166, Fukuoka
  - 187, Fukushima
  - 107, Gifu
  - 162, Himeji
  - 110, Hiroshima
  - 117, Hokkaido
  - 130, Hokkaido
  - 176, Hokkaido
  - 143, Kagoshima
  - 156, Kagoshima
  - 120, Kodaira
  - 105, Kokubunji
  - 306, Kōshi
  - 172, Miyazaki
  - 179, Miyazaki
  - 305, Nagoya
  - 106, Niigata
  - 153, Niigata
  - 109, Okayama
  - 174, Osaka
  - 119, Saitama
  - 147, Sakai
  - 194, Sakai
  - 304, Sapporo
  - 138, Tochigi
  - 184, Tokyo
  - 190, Tokyo
  - 111, Ube

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in Japan in June 2011.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS) which consisted of all subjects who took at least one dose of study medication in this study.
Groups:
- Levetiracetam: Levetiracetam dose was be adjusted at the investigator's discretion in the range from 20mg/kg/day or 1000mg/day to 60mg/kg/day or 3000mg/day during this study
Period: Overall Study
Arm/Group | Levetiracetam
Started | 44
Completed | 34
Not Completed | 10
Not completed — Withdrawal by Subject | 4
Not completed — AE, non-serious non-fatal | 4
Not completed — Withdrawal Criteria No.3 | 1
Not completed — Subject moved a long distance | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Safety Set (SS) which consisted of all subjects who took at least one dose of study medication in this study.
Arm/Group | Levetiracetam
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 Years | 28
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events During the Entire Study Period
Time Frame: Through study completion, an average of 3 years
Population: The Safety Set (SS) consisted of all subjects who took at least one dose of study medication in this study.
Measure: Number; unit: Treatment Emergent Adverse Events
Groups:
- Levetiracetam (SS): Levetiracetam dose was be adjusted at the investigator's discretion in the range from 20mg/kg/day or 1000mg/day to 60mg/kg/day or 3000mg/day during this study
Arm/Group | Levetiracetam (SS)
Number analyzed (Participants) | 44
Treatment Emergent Adverse Events | 626

2. Secondary Outcome: The Percentage Change in Generalized Tonic-Clonic (GTC) Seizure Frequency Per Week Over the Evaluation Period From Either of the Combined Baseline Periods of the Previous Studies (N01159 or N01363).
Description: Percentage change in generalized tonic-clonic (GTC) seizure frequency per week from Baseline of previous studies B over the Treatment Period A is calculated using the equation:
  Percentage change from Baseline = ((A-B)/B)*100. Percentage change from baseline is not defined for subjects whose baseline information is missing / unknown or equal to zero, or whose seizure frequency per week is missing/unknown. A negative value in change in generalized tonic-clonic (GTC) seizure frequency indicates a reduction of generalized tonic-clonic (GTC) seizure frequency over the Treatment Period.
Time Frame: During the Treatment Period (up to 4.8 years)
Population: The Full Analysis Set (FAS) consisted of all subjects with evaluable baseline and post-baseline values of generalized tonic-clonic (GTC) seizure frequency as the efficacy analysis, excluding those patients who seriously violated Good Clinical Practice (GCP).
Measure: Median (95% Confidence Interval); unit: percent change
Groups:
- Levetiracetam (FAS): Levetiracetam dose was be adjusted at the investigator's discretion in the range from 20mg/kg/day or 1000mg/day to 60mg/kg/day or 3000mg/day during this study
Arm/Group | Levetiracetam (FAS)
Number analyzed (Participants) | 43
percent change | -92.07 [-97.16 to -64.64]

3. Secondary Outcome: The Incidence of Adverse Drug Reactions During the Entire Study Period
Description: Adverse drug reactions excludes Adverse Events (AEs) described by the investigators with no relationship to study drug.
Time Frame: Through study completion, an average of 3 years
Population: The Safety Set (SS) consisted of all subjects who took at least one dose of study medication in this study.
Measure: Number; unit: Adverse Drug Reactions
Arm/Group | Levetiracetam (SS)
Number analyzed (Participants) | 44
Adverse Drug Reactions | 46

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Visit 1 (Week 0) until Safety Follow Up Visit (up to 4.7 years).
Description: Advers events refers to the Safety Set (SS) which consisted of all subjects who took at least one dose of study medication in this study.
Arm/Group | Levetiracetam (SS)
Serious Adverse Events (participants affected / at risk) | 13/44
Other Adverse Events (participants affected / at risk) | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (SS) (N=44)
Influenza (Infections and infestations) | 2 (2)
Acute tonsillitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Medical observation (Investigations) | 1 (1)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (7)
Breast adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Abortion induced (Surgical and medical procedures) | 1 (1)
Scoliosis surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (SS) (N=44)
Dental caries (Gastrointestinal disorders) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 8 (14)
Constipation (Gastrointestinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 4 (5)
Pyrexia (General disorders) | 8 (14)
Nasopharyngitis (Infections and infestations) | 35 (138)
Influenza (Infections and infestations) | 9 (12)
Otitis media (Infections and infestations) | 6 (6)
Gastroenteritis (Infections and infestations) | 5 (11)
Bronchitis (Infections and infestations) | 3 (5)
Conjunctivitis (Infections and infestations) | 3 (3)
Pulpitis dental (Infections and infestations) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 7 (16)
Excoriation (Injury, poisoning and procedural complications) | 6 (32)
Wound (Injury, poisoning and procedural complications) | 4 (4)
Weight increased (Investigations) | 5 (6)
Electrocardiogram QT prolonged (Investigations) | 3 (3)
Protein urine present (Investigations) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Convulsion (Nervous system disorders) | 16 (40)
Somnolence (Nervous system disorders) | 10 (10)
Headache (Nervous system disorders) | 9 (21)
Dizziness (Nervous system disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 5 (6)
Skin erosion (Skin and subcutaneous tissue disorders) | 4 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days